CLINICAL TRIAL: NCT00349050
Title: Transcranial Magnetic Stimulation (TMS) Effects on Pain Perception
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: K23NS050485-01A2 (NIH); K23NS050485-01A2 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2010-10

CONDITIONS: Pain; Trigeminal Neuralgia; Neuropathic Pain
Keywords: trigeminal neuralgia; neuropathic pain; complex regional pain syndrome; reflex sympathetic dystrophy; pain; chronic pain; transcranial magnetic stimulation; TMS; laboratory pain assessment
MeSH Terms: conditions — Pain; Trigeminal Neuralgia; Neuralgia; Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy; Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): laboratory pain assessment
  Interventions: Device: laboratory pain assessment
- 2 (Active Comparator): transcranial magnetic stimulation
  Interventions: Procedure: transcranial magnetic stimulation

INTERVENTIONS:
Device: laboratory pain assessment — Participants will record their pain experiences every day for 2 weeks before receiving the first of 5 laboratory pain assessments. The laboratory pain assessment uses a small device, controlled by a computer and attached to the underside of the forearm, to produce different temperature stimulations. As the device reaches a level considered painful to the participant, he/she can push a button to return to a level of comfort.
  Arms: 1
Procedure: transcranial magnetic stimulation — There will be two, 20-minute, 3-day TMS treatment sessions. Participants will be randomly assigned to one of two groups. Group A will receive real TMS for the first 3-day treatment and "sham" TMS (which does not involve real stimulation) for the second treatment. Group B will receive "sham" TMS for the first treatment, and real TMS for the second treatment. Regardless of the group, participants will receive both real and "sham" TMS.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effects of transcranial magnetic stimulation on pain perception.

DETAILED DESCRIPTION:
Chronic pain represents a huge public health concern and is generally poorly understood at a basic neurobiological level. Transcranial magnetic stimulation (TMS) is a non-invasive technique that uses electromagnetic pulses to temporarily stimulate specific brain areas in awake people (without the need for surgery, anesthesia, or other invasive procedures). Previous research suggests that TMS may be effective in reducing pain perception in healthy adults and in patients with various types of pain conditions, such as neuropathic pain. However, there is relatively little research on TMS and pain that addresses optimal TMS device parameters, optimal cortical targets, and potential differences in response to TMS between healthy persons and those with chronic pain.

The purpose of this trial is to study the effects of TMS on pain perception. Specifically, this study will determine optimal device parameters (dose) and brain targets for stimulation with TMS in order to reduce pain in patients with neuropathic pain and in healthy adults using laboratory pain methods.

Participants with Neuropathic Pain:

After an initial screening, eligible participants with neuropathic pain will receive a magnetic resonance imaging (MRI) scan to help determine the best target for TMS stimulation later in the study. Participants will be asked to record their pain experiences every day for 2-4 weeks before receiving the first of 2 laboratory pain assessments. The laboratory pain assessment uses a small device, controlled by a computer and attached to the underside of the forearm, to produce different temperature stimulations. As the device reaches a level considered painful to the participant, he/she can push a button to return to a level of comfort.

The next part of the trial involves two, 20-minute TMS treatment sessions per day for 5-days. Participants will be randomly assigned to one of two groups. Group A will receive real TMS and Group B will receive "sham" TMS. Study participation time for individuals with TGN is about 8 weeks, including about 10 hours (7 visits) at the Medical University of South Carolina (MUSC).

Healthy Volunteers:

In addition to an interview with researchers regarding medical history, healthy participants will complete a self-report screening to assess pain history and level of depression and anxiety. Eligible participants will be given a laboratory pain assessment, and be randomly assigned to one of two groups: group A will receive real TMS and group B will receive "sham" TMS. After TMS, participants will receive another full laboratory pain assessment and complete questionnaires. For healthy volunteers, participation in the study will take about 3 hours and may be completed in one or two visits.

ELIGIBILITY:
Inclusion Criteria:

For Healthy Adults:

* Between age of 21 and 60
* No prescription medications in previous 3 months
* No seizure history
* No depression
* Not suicidal
* No anxiety
* No hospitalizations or surgeries in previous 6 months
* No history of chronic pain conditions
* No implanted metal devices (e.g., pacemakers, metal plates, wires)
* Not pregnant
* No alcohol abuse/dependence history in previous 6 months
* No illicit drug use in previous 6 months
* Capable of reading, writing, giving consent, following instructions
* No history of brain surgery or history of loss of consciousness >15 minutes
* No history of autoimmune or endocrine disorder
* No significant anxiety about entering MRI scanner

For Patients with neuropathic pain:

* Between age of 21 and 75
* No seizure history
* Not taking medications shown to increase seizure risk (6 months)
* Not suicidal
* No hospitalizations or surgeries in previous 3 months
* No implanted metal devices (e.g., pacemakers, metal plates, wires)
* Not pregnant
* No alcohol abuse/dependence history in previous 6 months
* No illicit drug use in previous 6 months
* Capable of reading, writing, giving consent, following instructions
* Chronic pain (>6 months), not significantly relieved by pharmacological treatment
* No significant anxiety about entering MRI scanner

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Clinical neuropathic pain ratings, activity levels, analgesic medication usage, mood ratings, laboratory pain measures (thermal and mechanical pain thresholds, suprathreshold pain ratings, and wind-up pain ratings). | measured during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Borckardt, Ph.D., Principal Investigator — Department of Psychiatry and Behavioral Sciences, Medical University of South Carolina
Locations (1):
- Brain Stimulation Laboratory, Department of Psychiatry and Behavioral Sciences Medical University of South Carolina 5-North, IOP, 67 President Street, Charleston, South Carolina, United States